CLINICAL TRIAL: NCT03956628
Title: Evaluation of Preventive (Stay Safe) Training Program of Child Abuse for Teachers and Children: A Randomized Controlled Trial From Multan City
Brief Title: Evaluation of Preventive (Stay Safe) Training Program of Child Abuse for Teachers and Children
Acronym: intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahauddin Zakariya University (Other)
Responsible Party: Principal Investigator, Zainab noor Hussain, Principal investigator, Bahauddin Zakariya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MPP-17-07
Record Dates: First submitted 2019-05-03; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Child Abuse

STUDY DESIGN:
Intervention Model Description: There are two groups, experimental and control group. Experimental group will be provided with psycho education about safety skills related to child abuse. Control group will not be given any intervention.
Who Masked: Participant
Masking Description: Participants are randomly assigned to control and experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): participants in experimental group receive intervention and experimental group consists of two sub groups, teachers and students.
  Interventions: Behavioral: stay safe program
- control group (No Intervention): participants in control group does not receive intervention and control group consists of two sub groups, teachers and students.

INTERVENTIONS:
Behavioral: stay safe program — Prevention consist of 5-6 lessons having topics about learning safety skills which includes identifying touch, safe and unsafe environment/events, bullying, the good or bad secrets and strangers.
  Arms: experimental group

SUMMARY:
The current study aims to elaborate the effectiveness of stay safe programme which is a child abuse prevention programme for children, this study examine the effectiveness of this programme on children and teachers of Multan city schools. Mainly, this study enhance the understanding of teachers and children to provide protection and confidence by following programme.

DETAILED DESCRIPTION:
The study examine the stay safe programme effectiveness among school teachers and children, as Pakistan is today badly indulge in this issue; In this circumstances this type of study provide essential role in society. some schools from Multan city are included, the quasi experimental study is used, where the participants are randomly divided into two groups (control and experimental). school based sampling method is used where different campuses of one school is included, through random number generator, six schools are selected for participation where 3 schools are included in control group and 3 are in experimental group. the participants consist of school teachers and children, where each group (children & teachers) is further divided into control and experimental group. children and teachers of class 1 and 2 are included. scales used in the study are Battle self-esteem inventory and children knowledge and skills questionnaire for children while teachers knowledge and skills questionnaire for teachers is used in study. 1 week time gap is also considered between pre and post testing for better examination of change. stay safe programme is very powerful tool as it cover different sensitive issues and provide confidence or safety skills to children.it also provide teachers with the strategies that they should use to make classroom environment healthy or encourage children to speak up and also provide guidance to deal with issues safely and listen every child carefully. Different videos, worksheets, basic knowledge that cover 5 major topics like feeling safe and unsafe, wanted and unwanted touch, bullying, tell adults about negative interaction with bullies and victimizers, strangers and dealing with strangers are all include in the stay safe programme. The lessons that include in this programme are so healthy and best for the protection of child, it also boost their self-esteem and make them worthy and active cognitively. informed consent is provided to participants for initiating the study properly, as it is ethical. every participant data would be confidential or the theme of study would be debrief to the control group after study.

ELIGIBILITY:
Inclusion Criteria:

1. students enrolled in class 1-2
2. age range between 5-9
3. students allowed by their parents to participate in the study.

Exclusion Criteria:

1. students not enrolled in class 1 or 2
2. students not within age range.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 378 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Children Safety Knowledge and Skills Questionnaire (SKSQ) | 2 months
  the scale consist of 18 items. it is an open ended questionnaire which consist of the scoring key is 4- someone you don't know, 3- man/woman you don't know, 2- no response or don't know and 1- misconception.It measure the knowledge of children about strangers, bullying, touch, secrets, lost, disclosure and bribes. these are the sub scales and sub scales sum up to make a total score for each child. the items of scale deal with different knowledge and skills of children related to self-protection. The range of scoring is from 18 to 80 for complete questionnaire.maximum value is 80 and minimum is 18. Internal consistency reliability coefficient in regards to the stay safe programme (alpha = .79). if a child get 18 scores that means his safety knowledge is low while 80 means knowledge is high. this score obtains after sum up or average of the total sub scales.
Teachers' Knowledge/Attitudes Questionnaire (TKAQ) | 2 months
  A 38 item questionnaire which assessed knowledge of prevalence, causes and indicators of child sexual abuse as well as characteristics of victims and offenders. In addition it examined parents' self-reports of the likelihood of them believing a child's disclosure of abuse, attributions of responsibility for sexual victimisation attitudes towards prevention, knowledge of and attitudes towards services and confidence/anxieties relating to sexual abuse.
  Parents responded to each item on a five point Likert scale ranging from "strongly agree" to "strongly disagree". For 22 items "strongly agree" is the correct response and for 16 items "strongly disagree" is correct. Each item is scored from 1 to 5 and the potential range for total scores is from 38 to 190. The alpha co-efficient for the total questionnaire was .80, indicating good internal consistency reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Rizwana Amin, PhD, Principal Investigator — Bahauddin Zakariya University Multan
Locations (1):
- Zainab noor Hussain, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacIntyre D, Carr A. Evaluation of the effectiveness of the stay safe primary prevention programme for child sexual abuse. Child Abuse Negl. 1999 Dec;23(12):1307-25. doi: 10.1016/s0145-2134(99)00092-7. PMID 10626613
- [Result] MacIntyre D, Carr A. Helping children to the other side of silence: a study of the impact of the stay safe programme on Irish children's disclosures of sexual victimization. Child Abuse Negl. 1999 Dec;23(12):1327-40. doi: 10.1016/s0145-2134(99)00097-6. PMID 10626614
- See also: this article was cited in the study — https://www.ncbi.nlm.nih.gov/pubmed/10626613
- Available data/document: stay safe programme — http://www.staysafe.ie — data can be accessed by approaching the above specified cite as it has programme that was used in the study.

DOCUMENTS (3):
  • Informed Consent Form (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03956628/ICF_000.pdf
  • Study Protocol (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03956628/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03956628/SAP_002.pdf